CLINICAL TRIAL: NCT03762460
Title: Pilot Randomized Clinical Trial of eHealth Tools
Brief Title: A Pilot Study of eHealth Tools in a Tertiary-care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other); Healthy Minds Canada (Unknown); Pfizer (Industry)
Responsible Party: Principal Investigator, Raymond Lam, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H17-02786; V17-02786 (Other: Vancouver Coastal Health Research Institute)
Record Dates: First submitted 2018-04-11; First posted 2018-12-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Depression
Keywords: Measurement-Based Care; e-Mental Health; Functional Outcomes; Occupational Functioning; Cognition; Mobile Technology
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online eHealth Tool (Experimental): Participants randomized to this group will use a personally-owned smartphone, tablet, or computer to access the online eHealth tool.
  Interventions: Other: Online eHealth tool
- Informational website (control) (Placebo Comparator): Participants randomized to this group will receive information about online resources for mental health
  Interventions: Other: Informational website

INTERVENTIONS:
Other: Online eHealth tool — Mobile-optimized online eHealth tool to support MBC.
  Arms: Online eHealth Tool
Other: Informational website — Participants randomized to this group will receive information about online resources for mental health
  Arms: Informational website (control)

SUMMARY:
This feasibility study investigates the use of eHealth tools within routine medical treatment for patients with depression in an outpatient psychiatric setting. The study investigates whether patients find a mobile-optimized online eHealth tool to be acceptable and feasible, and whether clinical and functional outcomes improve with use of the online eHealth tool, compared to informational online resources for mental health.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is increasingly recognized as the most common psychiatric disorder and as one of the most common medical diagnoses worldwide.

Measurement-based care (MBC) is an evidence-based approach for providing effective clinical care to patients with MDD. MBC utilizes validated rating scales to assess symptom severity, functional impairments, treatment adherence, and side-effect burden to personalize clinical decision-making based on measured outcomes and clinical algorithms. However, despite evidence demonstrating improved outcomes, MBC is still not routinely used by physicians. Barriers to the use of MBC include lack of knowledge of which scales to use, how to incorporate measurements into clinical charting systems, and the extra time needed for repeated assessments.

Our research team developed a web-based application (app) optimized for mobile devices to address the treatment gap in MBC for people with depression, especially those who are working while depressed. This user-friendly eHealth tool encourages patients to actively participate in MBC by using their smartphones, tablets, or computers to screen, monitor, and manage depressive symptoms and functional outcomes. Results can be easily displayed and printed to share with clinicians, thereby affording health professionals a simple and cost-effective means to integrate MBC into standard practices and to optimize treatment for MDD at the point of care, without needing additional materials, equipment, or staffing.

This research study investigates the feasibility of using a mobile-optimized online eHealth tool to support MBC in routine clinical care for MDD within an outpatient psychiatric setting.

To determine both the clinical and practical utility of eMBC, this study will enroll "real-world" patients with few exclusion criteria and undergoing naturalistic treatments so that findings will be generalizable to other clinical settings and practices.

Note: As of April, 2020 (before recruitment started), because of the pandemic the study protocol was changed to be fully virtual, with a change in the primary outcome to a patient feasibility outcome.

ELIGIBILITY:
Inclusion Criteria:

1. age 19-65 and capable of informed consent;
2. diagnosis of major depressive episode (MDE) by the Diagnostic and Statistical Manual, Fifth Edition (DSM-5) criteria as determined by the clinic psychiatrist;
3. at least moderate depression as defined by QIDS-SR score of 10 or higher on the Quick Inventory for Depressive Symptomatology, Self-Rated (QIDS-SR);
4. access to an Internet-enabled computer or mobile device; and
5. able to read and understand English sufficiently to use the eMBC platform

Exclusion Criteria:

1. active psychotic or substance use disorder; or
2. severe suicidality as judged by the psychiatrist.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility-of-use outcome: Percentage of patients who use the eHealth tool (MoodFx) 3 or more times over the 6-month period | 6 months
  Percentage of patients who use the eHealth tool (MoodFx), defined as 3 or more uses over the 6-month follow up period

SECONDARY OUTCOMES:
Change scores on the Quick Inventory of Depressive Symptomatology (QIDS-SR) from baseline to follow up at 8 weeks and 6 months. | 8 weeks and 6 months
  The Quick Inventory of Depressive Symptomatology (QIDS-SR) is a self-report scale to assess symptoms of depression and consists of 16 items, 9 of which contribute to a summed total score (i.e., only the highest score of items 1-4, 6-9, and 15-16 are counted towards the total score). Higher scores indicate more severe symptoms, with individual item scores ranging from 0-3 and total scores ranging from 0-27.
Change scores on the Patient Health Questionnaire (PHQ-9) from baseline to follow up at 8 weeks and 6 months. | 8 weeks and 6 months
  The Patient Health Questionnaire (PHQ-9) is a brief, self-rated scale assessing symptoms of depression. The scale consists of 9 items rated on a scale from 0-3, with higher scores indicating more severe symptoms. Item scores are summed to yield a total score, range 0-27.
Change scores on the Generalized Anxiety Disorder scale (GAD-7) from baseline to follow up at 8 weeks and 6 months. | 8 weeks and 6 months
  The Generalized Anxiety Disorder scale (GAD-7) is a brief, self-rated scale assessing symptoms of generalized anxiety. The scale consists of 7 items rated on a scale from 0-3, with higher scores indicating more severe symptoms. Item scores are summed to yield a total score, range 0-21.
Change scores on the Sheehan Disability Scale (SDS) from baseline to follow up at 8 weeks and 6 months. | 8 weeks and 6 months
  The Sheehan Disability Scale (SDS) is a brief self-report scale assessing functional impairment in three inter-related domains: work/school, social and home/family life. The user rates the extent to which work/school, social life and home life or family responsibilities are impaired by his or her symptoms on a 11 point visual analog scale (range 0-10). Higher scores indicate greater impairment.
Change scores on the Lam Employment Absence and Productivity Scale (LEAPS) from baseline to follow up at 8 weeks and 6 months. | 8 weeks and 6 months
  The Lam Employment Absence and Productivity Scale (LEAPS) is a brief self-rated scale to assess patients' work functioning. The LEAPS consists of 10 items rated on a 5-point scale from 0-4, with higher scores indicating greater impairment. Item scores are summed to yield a total score, range 0-28.
Change scores on the Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF) from baseline to follow up at 8 weeks and 6 months. | 8 weeks and 6 months
  The Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) is a 16 item self-administered questionnaire assessing life satisfaction over the past week. Each question is rated on a 5 point scale from 1 (Very Poor) to 5 (Very Good). Scores from the individual items are added together and reported as percentage maximum possible score.
Change scores on the Euro-QOL-5Lscale (EQ-5D-5L) from baseline to follow up at 8 weeks and 6 months. | 8 weeks and 6 months
  The Euro-QOL scale (EQ-5D) is a standardised self-report instrument for measuring generic health status. It consists of 5 items evaluating rated on a 5-level scale from no impairments to complete impairment. The 5 rating levels can be quantified as ranging from 0 to 4, with higher scores indicating higher impairment. Total score ranges from 0 to 20.
Satisfaction with eHealth tool as measured by the System Usability Scale. | 6 months
  The System Usability Scale is a 10-item survey that evaluates user satisfaction with online tools, applications, etc. Each item is rated on a 5-point scale (from 0-4), with higher scores indicating greater satisfaction. Item scores may be added together to yield scores ranging from 0-40, and then multiplied by 2.5 for scores ranging from 0-100. (Note these scores are not percentages or percentiles.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond W Lam, MD, Principal Investigator — University of British Columbia
Locations (1):
- UBC Mood Disorders Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No